CLINICAL TRIAL: NCT04563988
Title: Factors for Predicting Severe Asthma Exacerbators in Adult Asthmatics: A Real Word- Effectiveness Study
Status: Completed | Type: Observational
Sponsor: Hae-Sim Park (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Hae-Sim Park, Principal investigator, Clinical professor, Department of Allergy and Clinical Immunology, Ajou University School of Medicine
Organization: Ajou University School of Medicine (Other)
Other Study IDs: AJIRB-MED-MDB-18-291
Record Dates: First submitted 2020-08-31; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-center, retrospective, cross-sectional study. It plan to investigate the predictors for asthma exacerbation in long term follow up real world management with analyzing big data of electronic medical records (EMR).

DETAILED DESCRIPTION:
The long-term goals of asthma treatment are to achieve well control of symptoms and to minimize the future risk of asthma exacerbations (AEs). Asthma is a heterogeneous disease with various responses to treatment and clinical outcomes. AEs are a prominent feature of severe asthmatics; however, frequent AEs have also been reported in mild asthmatics.

This is a prospectively designed observational study to identify predictors for patients with frequent AEs among adult asthmatics by analyzing medical big data of electronic medical records (EMR), which will provide an insight in the long-term management of adult asthmatics in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥17 years
* Patients having bronchial asthma with J45-J46 code of International classification of Diseases (10th edition on EMR)
* Asthmatics who had been treated by allergy or respiratory specialists

Exclusion Criteria:

* Patients who has less than one year for asthma treatment

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged ≥17 years diagnosed as having bronchial asthma (with J45-J46 code of International classification of Diseases, 10th edition on EMR) and who had been treated by allergy or respiratory specialists at Ajou University Hospital from January 1995 to June 2018
Sampling Method: Non-Probability Sample
Enrollment: 5058 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Identifying prognostic factors for risk of severe asthma exacerbation | During the initial 2 years
  Identifying prognostic factors for risk of severe asthma exacerbation

SECONDARY OUTCOMES:
Evaluating total IgE (KU/L) to predict severe asthma exacerbation | During 10 years of treatment
  Evaluating total IgE (KU/L) to predict severe asthma exacerbation
Evaluating peripheral eosiniphil, neutrophil, basophil and lymphocyte counts to predict severe asthma exacerbation | During 10 years of treatment
  Unit of peripheral eosiniphil, neutrophil, basophil and lymphocyte counts: ×10³/uL
Evaluating ECP (ug/L) to predict severe asthma exacerbation | During 10 years of treatment
  Evaluating ECP (ug/L) to predict severe asthma exacerbation
Evaluating sputum eosinophils (%) to predict severe asthma exacerbation | During 10 years of treatment
  Evaluating sputum eosinophils (%) to predict severe asthma exacerbation
Evaluating FEV1 (%) and FEV1/FVC (%) to predict severe asthma exacerbation | During 10 years of treatment
  Evaluating FEV1 (%) and FEV1/FVC (%) to predict severe asthma exacerbation
Comparing clinical characteristics according to the frequency of severe asthma exacerbation | During the initial 2 years
  Comparing clinical characteristics according to the frequency of severe asthma exacerbation
Sensitivity and specificity of predictors | during the initial 2 years and the following 3-10 years of treatment
  Sensitivity and specificity of predictors

CONTACTS AND LOCATIONS:
Overall Officials: Hae-sim Park, MD, PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Greenberg S. Asthma exacerbations: predisposing factors and prediction rules. Curr Opin Allergy Clin Immunol. 2013 Jun;13(3):225-36. doi: 10.1097/ACI.0b013e32836096de. PMID 23635528
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] van Veen IH, Ten Brinke A, Sterk PJ, Sont JK, Gauw SA, Rabe KF, Bel EH. Exhaled nitric oxide predicts lung function decline in difficult-to-treat asthma. Eur Respir J. 2008 Aug;32(2):344-9. doi: 10.1183/09031936.00135907. Epub 2008 May 28. PMID 18508818
- [Background] Bayes HK, Cowan DC. Biomarkers and asthma management: an update. Curr Opin Allergy Clin Immunol. 2016 Jun;16(3):210-7. doi: 10.1097/ACI.0000000000000263. PMID 27057795
- [Background] Parulekar AD, Diamant Z, Hanania NA. Role of T2 inflammation biomarkers in severe asthma. Curr Opin Pulm Med. 2016 Jan;22(1):59-68. doi: 10.1097/MCP.0000000000000231. PMID 26574724
- [Background] Buhl R, Korn S, Menzies-Gow A, Aubier M, Chapman KR, Canonica GW, Picado C, Martin N, Escobar RA, Korom S, Hanania NA. Assessing biomarkers in a real-world severe asthma study (ARIETTA). Respir Med. 2016 Jun;115:7-12. doi: 10.1016/j.rmed.2016.04.001. Epub 2016 Apr 14. PMID 27215497
- [Background] Humbert M, Busse W, Hanania NA, Lowe PJ, Canvin J, Erpenbeck VJ, Holgate S. Omalizumab in asthma: an update on recent developments. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):525-36.e1. doi: 10.1016/j.jaip.2014.03.010. Epub 2014 Jun 11. PMID 25213045
- [Background] Grimaldi-Bensouda L, Zureik M, Aubier M, Humbert M, Levy J, Benichou J, Molimard M, Abenhaim L; Pharmacoepidemiology of Asthma and Xolair (PAX) Study Group. Does omalizumab make a difference to the real-life treatment of asthma exacerbations?: Results from a large cohort of patients with severe uncontrolled asthma. Chest. 2013 Feb 1;143(2):398-405. doi: 10.1378/chest.12-1372. PMID 23505637
- [Background] Zissler UM, Esser-von Bieren J, Jakwerth CA, Chaker AM, Schmidt-Weber CB. Current and future biomarkers in allergic asthma. Allergy. 2016 Apr;71(4):475-94. doi: 10.1111/all.12828. Epub 2016 Jan 18. PMID 26706728